CLINICAL TRIAL: NCT02789709
Title: Metabolomic Phenotyping After Surgery for Colon Cancer: Study of Novel Predictive Biomarkers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Collaborators: University of Barcelona (Other)
Responsible Party: Principal Investigator, Miguel Pera, MD, Parc de Salut Mar
Other Study IDs: PI15/00458
Record Dates: First submitted 2016-05-30; First posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non metastatic colon cancer patients: Consecutive patients undergoing elective surgery for non-metastatic colon or rectal cancer with curative intent.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Segmental resection for colon cancer and anterior resection in patients with rectal cancer

SUMMARY:
Predictive biomarkers are needed to identify those patients with higher risk of recurrence after surgery for colon cancer with curative intent. Our main objective is to determine a metabolite profile in blood plasma from patients operated from colorectal cancer that can be associated with the oncologic outcome and be validated as predictive biomarkers in future studies. A secondary objective is to study the glycolytic metabolism of colon cancer cell lines treated with plasma samples from the same patients. In particular, to validate the increased utilization of lactate by tumor cells as a metabolic substrate using postoperative human samples.

Patients with colorectal cancer that have undergone surgical resection will be included. Plasma samples will be obtained before surgery and the 4th day and the 3rd, 6th, 12th, and 18th months after surgery. Metabolic profiles in plasma samples will be determined using a kit that allows the quantification of 180 metabolites by mass spectrometry.

A clinical follow up will be maintained for at least 2 years to identify tumor recurrences.

DETAILED DESCRIPTION:
Up to 30-40% of patients operated from colorectal cancer display tumor recurrence. Predictive biomarkers are needed to identify those patients with higher risk of recurrence. Our main objective is to determine a metabolite profile in blood plasma from patients operated from colorectal cancer that can be associated with the oncologic outcome and be validated as prognostic biomarkers in future studies. A secondary objective is to study the glycolytic metabolism of colon cancer cell lines treated with plasma samples from the same patients. In particular, to validate the increased utilization of lactate by tumor cells as a metabolic substrate using postoperative human samples, as it was previously observed by us in vitro using an inflammatory environment in conditions of hypoxia and lack of glucose. Patients with colorectal cancer that have undergone surgical resection will be included. Plasma samples will be obtained before surgery and the 4th day and the 3rd, 6th, 12th, and 18th months after surgery. Metabolic profiles in plasma samples will be determined using a kit that allows the quantification of 180 metabolites by mass spectrometry. Cellular assays will be performed on the SW620 and HT-29 colon cancer cell lines. Cells will be treated with plasma samples and the concentration of lactate and other metabolites will be analyzed in the medium supernatants. A clinical follow up will be maintained for at least 2 years to identify tumor recurrences.

ELIGIBILITY:
Inclusion Criteria:

* Non-metastatic colon and rectal cancer undergoing surgery with curative intent
* Patients signed informed consent

Exclusion Criteria:

* Patients undergoing preoperative chemotherapy and/or radiotherapy
* Emergency surgery
* Surgical resection R1 or R2
* Patients presenting with other known malignancies for which they are receiving treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing surgery for colon and rectal cancer with curative intent
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 5 years from the date of surgery
  Time from the date of surgery to the date of first documentation of recurrence

SECONDARY OUTCOMES:
Disease-specific survival | 5 years from the date of surgery
  Time from the date of surgery to death by colon cancer
Local recurrence | 5 years from the date of surgery
  Tumor associated with surgical site (anastomosis, tumor bed, and mesentery) and confirmed histologically or by imaging.
Systemic recurrence | 5 years from the date of surgery
  Spread of the disease outside the surgical field to organs such as the liver, lungs, bones, or brain
Postoperative intra-abdominal sepsis | 30 days from the date of surgery
  Anastomotic leak or intra-abdominal abscess
Postoperative mortality | 30 days from the date of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar Medical Research Institute, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pera M, Nelson H, Rajkumar SV, Young-Fadok TM, Burgart LJ. Influence of postoperative acute-phase response on angiogenesis and tumor growth: open vs. laparoscopic-assisted surgery in mice. J Gastrointest Surg. 2003 Sep-Oct;7(6):783-90. doi: 10.1016/s1091-255x(03)00111-2. PMID 13129557
- [Result] Bohle B, Pera M, Pascual M, Alonso S, Mayol X, Salvado M, Schmidt J, Grande L. Postoperative intra-abdominal infection increases angiogenesis and tumor recurrence after surgical excision of colon cancer in mice. Surgery. 2010 Jan;147(1):120-6. doi: 10.1016/j.surg.2009.06.035. Epub 2009 Sep 20. PMID 19767043
- [Result] Pascual M, Alonso S, Pares D, Courtier R, Gil MJ, Grande L, Pera M. Randomized clinical trial comparing inflammatory and angiogenic response after open versus laparoscopic curative resection for colonic cancer. Br J Surg. 2011 Jan;98(1):50-9. doi: 10.1002/bjs.7258. Epub 2010 Aug 26. PMID 20799296
- [Result] Pascual M, Bohle B, Alonso S, Mayol X, Salvans S, Grande L, Pera M. Preoperative administration of erythropoietin stimulates tumor recurrence after surgical excision of colon cancer in mice by a vascular endothelial growth factor-independent mechanism. J Surg Res. 2013 Jul;183(1):270-7. doi: 10.1016/j.jss.2012.12.041. Epub 2013 Jan 16. PMID 23348072
- [Result] Salvans S, Mayol X, Alonso S, Messeguer R, Pascual M, Mojal S, Grande L, Pera M. Postoperative peritoneal infection enhances migration and invasion capacities of tumor cells in vitro: an insight into the association between anastomotic leak and recurrence after surgery for colorectal cancer. Ann Surg. 2014 Nov;260(5):939-43; discussion 943-4. doi: 10.1097/SLA.0000000000000958. PMID 25243554
- [Result] Espin E, Ciga MA, Pera M, Ortiz H; Spanish Rectal Cancer Project. Oncological outcome following anastomotic leak in rectal surgery. Br J Surg. 2015 Mar;102(4):416-22. doi: 10.1002/bjs.9748. Epub 2015 Jan 26. PMID 25619499
- [Result] Alonso S, Pascual M, Salvans S, Mayol X, Mojal S, Gil MJ, Grande L, Pera M. Postoperative intra-abdominal infection and colorectal cancer recurrence: a prospective matched cohort study of inflammatory and angiogenic responses as mechanisms involved in this association. Eur J Surg Oncol. 2015 Feb;41(2):208-14. doi: 10.1016/j.ejso.2014.10.052. Epub 2014 Nov 1. PMID 25468742
- [Derived] Montcusi B, Madrid-Gambin F, Pozo OJ, Marco S, Marin S, Mayol X, Pascual M, Alonso S, Salvans S, Jimenez-Toscano M, Cascante M, Pera M. Circulating metabolic markers after surgery identify patients at risk for severe postoperative complications: a prospective cohort study in colorectal cancer. Int J Surg. 2024 Mar 1;110(3):1493-1501. doi: 10.1097/JS9.0000000000000965. PMID 38116682